CLINICAL TRIAL: NCT05318027
Title: Use of Natural Language Processing ChatBot and Automated Continuous Activity Monitoring Via Mobile Phones for Early Detection and Management of Symptoms in Patients Undergoing Cancer Treatment
Brief Title: ChatBot and Activity Monitoring in Patients Undergoing Chemoradiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC 18921
Record Dates: First submitted 2021-12-06; First posted 2022-04-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Gastrointestinal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Monitoring and ChatBot (Experimental): Patients will receive standard of care chemotherapy and radiation therapy regimens, activity monitoring and utilize a ChatBot
  Interventions: Device: ChatBot
- Activity Monitoring without ChatBot (No Intervention): Patients will receive standard of care chemotherapy and radiation therapy regimens, activity monitoring alone

INTERVENTIONS:
Device: ChatBot — The automated chatbot will check in with the patient on two pre-specified days between scheduled outpatient visits. The chatbot will follow pre-specified symptom algorithms and classify symptoms as requiring high, intermediate and low risk follow ups. High risk symptoms will trigger a same day nursing/physician visit or telemedicine call/video. Intermediate risk symptoms will trigger a nursing triage visit or telemedicine call/video on the next day or treatment day. Low risk symptoms will notify the treating physician to address the symptoms at the next scheduled on treatment visit (OTV). If adjustments are needed in the chat bot triage algorithms, they will be updated in real time to decrease risk for adverse patient events.
  Arms: Activity Monitoring and ChatBot

SUMMARY:
Evaluate the feasibility of using a chatbot combined with continuous activity monitoring to proactively identify, appropriately triage and help manage patients' symptoms during cancer treatment Determine whether such an early outpatient clinic-based intervention can decrease rates of excess triage visits

Correlate changes in activity and early symptom management to emergency department visits, unplanned inpatient hospitalizations and treatment breaks

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >18 years) with a diagnosis of a head and neck, lung, gastrointestinal cancer, that are receiving concurrent chemotherapy and radiation treatment.
* Possession of a mobile device that can receive SMS texts and can deliver FitBit data wirelessly
* Ability read and respond in English
* Ability to provide informed consent to participate in the study

Exclusion Criteria:

* Patients who are bed bound at baseline (ECOG 4)
* Patients who rely on a wheelchair for ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of triage visits | 13 weeks
  Difference between Poisson event rates of triage visits between intervention and control arms

SECONDARY OUTCOMES:
Count of unplanned inpatient hospitalization | 13 weeks
Count of treatment breaks | 13 weeks
Count of emergency department visits | 13 weeks
Quality of Life scores | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arun Goel, MD, Principal Investigator — University of Pennsylvania; Kristine Kim, MD, Principal Investigator — University of Pennsylvania; Nishant Shah, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uyterlinde W. Overcoming toxicity-challenges in chemoradiation for non-small cell lung cancer. Transl Lung Cancer Res. 2016 Jun;5(3):239-43. doi: 10.21037/tlcr.2016.05.03. PMID 27413701
- [Background] Ghosh S, Rao PB, Kumar PR, Manam S. Concurrent Chemoradiation with Weekly Cisplatin for the Treatment of Head and Neck Cancers: an Institutional Study on Acute Toxicity and Response to Treatment. Asian Pac J Cancer Prev. 2015;16(16):7331-5. doi: 10.7314/apjcp.2015.16.16.7331. PMID 26514533
- [Background] Haj Mohammad N, Hulshof MC, Bergman JJ, Geijsen D, Wilmink JW, van Berge Henegouwen MI, van Laarhoven HW. Acute toxicity of definitive chemoradiation in patients with inoperable or irresectable esophageal carcinoma. BMC Cancer. 2014 Jan 31;14:56. doi: 10.1186/1471-2407-14-56. PMID 24485047
- [Background] Waddle MR, Chen RC, Arastu NH, Green RL, Jackson M, Qaqish BF, Camporeale J, Collichio FA, Marks LB. Unanticipated hospital admissions during or soon after radiation therapy: Incidence and predictive factors. Pract Radiat Oncol. 2015 May-Jun;5(3):e245-e253. doi: 10.1016/j.prro.2014.08.004. Epub 2014 Sep 17. PMID 25413398
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Lang K, Sussman M, Friedman M, Su J, Kan HJ, Mauro D, Tafesse E, Menzin J. Incidence and costs of treatment-related complications among patients with advanced squamous cell carcinoma of the head and neck. Arch Otolaryngol Head Neck Surg. 2009 Jun;135(6):582-8. doi: 10.1001/archoto.2009.46. PMID 19528407
- [Background] Beg MS, Gupta A, Stewart T, Rethorst CD. Promise of Wearable Physical Activity Monitors in Oncology Practice. J Oncol Pract. 2017 Feb;13(2):82-89. doi: 10.1200/JOP.2016.016857. PMID 28387544
- [Background] McNeely ML, Campbell KL, Rowe BH, Klassen TP, Mackey JR, Courneya KS. Effects of exercise on breast cancer patients and survivors: a systematic review and meta-analysis. CMAJ. 2006 Jul 4;175(1):34-41. doi: 10.1503/cmaj.051073. PMID 16818906